CLINICAL TRIAL: NCT01815476
Title: A Multicentre Randomized Controlled Clinical Trial for the Reduction of Acute Skin Reaction in Adjuvant Breast Radiation in Large Breasted Women Using a Prone Technique - The Prone Breast Trial
Brief Title: The Prone Breast Radiation Therapy Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Sunnybrook Regional Cancer Centre (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Danny Vesprini, MD, MSc, FRCPC, Radiation Oncologist, Toronto Sunnybrook Regional Cancer Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 380-2012
Record Dates: First submitted 2013-03-15; First posted 2013-03-21 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Ductal Carcinoma In Situ; Invasive Breast Cancer
Keywords: DCIS; Early Stage Invasive breast cancer; Prone breast radiotherapy
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT Positioning Intervention: Supine (Other): Patient will be treated in a supine position as per standard of care/control.
  Interventions: Radiation: Radiation Therapy Positioning Intervention
- RT Positioning Intervention: Prone (Experimental): Patient will be treated in the prone position.
  Interventions: Radiation: Radiation Therapy Positioning Intervention

INTERVENTIONS:
Radiation: Radiation Therapy Positioning Intervention — All participants will receive an adjuvant XRT dose to the breast of 50Gy in 25 fractions using an IMRT technique. In both arms, boost to the surgical bed using a mini-tangent technique will be delivered at the treating oncologist's discretion. Acceptable boost doses are 1600cGy/8 fractions, 1000cGy/5 fractions or 1325cGy/25 fractions as a simulatenous integrated boost. Participants randomized to the supine arm will be positioned supine on an angled breast board, with the ipsilateral arm abducted over her head. Participants randomized to the prone arm will be positioned prone on a prone breast board with both arms immobilized above the participant's head. The us of a cushion-like VaclocTM device is permitted at the treating physician's discretion. Radiation beams will be shaped to encompass the breast volume requiring treatment in both arms.

SUMMARY:
Participants undergoing radiation after breast conserving surgery for an early breast cancer (either Ductal Carcinoma In Situ (DCIS), or Early Stage Invasive breast cancer), and are at increased risk of developing a skin reaction because of their large breast size.

After breast conserving surgery (also known as a 'lumpectomy'), women with either DCIS or early stage invasive breast cancer receive radiation to the breast to decrease the risk of cancer recurrence. Breast radiation is usually done with women lying on their back ("supine"). Some women develop temporary breakdown of the skin (moist desquamation). This skin reaction can be painful and has been linked to long term side effects such as chronic pain and decreased quality of life.

This study is being done because women with large breasts have higher rates of skin breakdown (called 'moist desquamation') and breast pain during and shortly after radiation therapy is complete. It is unclear if such skin reactions and pain would be improved by alternating treatment position - namely lying on your belly ("prone") during their radiation treatment.

DETAILED DESCRIPTION:
The risk of moist desquamation in large breasted women remains unacceptably high and reactions tends to be severe and produce significant permanent and delayed side effects. Evidence suggests that the use of a prone breast IMRT technique has the potential to decrease the risk of moist desquamation in large breasted women to the levels that are now seen when average/smaller breasted women are treated with supine IMRT. As prone breast XRT is currently only offered at 6 of 15 of the Ontario Cancer Centres polled for the purposes of providing motivation for this study, a multicentre RCT is feasible to confirm and quantify the improvement provided by the prone technique and provide Level 1 evidence for it to be adopted world-wide.

ELIGIBILITY:
Inclusion Criteria:

* confirmed histological diagnosis of breast carcinoma or ductal carcinoma in situ (DCIS);
* treated with BCT;
* no indication for treatment of regional LN;
* Women with a bra size of 40 inches or greater, or a pre-surgery cup size of D or greater

Exclusion Criteria:

* Regional Lymph Node XRT indicated;
* Bilateral breast cancer;
* unhealed wound (skin not closed and/or infection);
* previous XRT to the same breast;
* unable to lie prone;
* presence of active connective tissue disease;
* pregnancy;
* unacceptable heart exposure (as measured by > 10% of the heart receiving 50% of the prescribed dose, i.e. V25Gy > 10%);
* adequate coverage of postoperative tumour bed not technically possible

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2013-05-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Moist Desquamation | 6-8 week post-treatment.
  Acute moist desquamation rates as measured by CTCAE 4.03 during and up to 6-8 weeks post treatment.

SECONDARY OUTCOMES:
Breast Pain | 6-8 week post-treatment.
  Acute breast pain rates as measured by CTCAE 4.03 and Visual Analog Scale (VAS) during and up to 6-8 weeks post treatment.
Radiation exposure of adjacent normal organs at risk | Day 1
  Determine if adjuvant breast IMRT in the prone position produces improved dose distribution in regards to exposure to critical structures including heart, lung, liver and contralateral breast when compared to treatment in the supine position.

OTHER OUTCOMES:
Patient Reported Quality of life | Questionnaires will be completed by subjects at time of radiation simulation as baseline, in the 5th week of radiation therapy treatment (during routine review) and at 6-8 week follow-up.
  Change in health related Quality of Life as per the EORTC core QoL questionnaire QLQ-C30 and the breast cancer module QLQ-BR23.

CONTACTS AND LOCATIONS:
Overall Officials: Danny Vesprini, MD MSc FRCPC, Principal Investigator — Toronto Sunnybrook Regional Cancer Centre
Locations (2):
- Canada (2):
  - British Columbia Cancer Agency - Vancouver Island centre, Victoria, British Columbia
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario

REFERENCES:
- [Derived] Vesprini D, Davidson M, Bosnic S, Truong P, Vallieres I, Fenkell L, Comsa D, El-Mallah M, Garcia L, Stevens C, Nakonechny K, Tran W, Kiss A, Rakovitch E, Pignol JP. Effect of Supine vs Prone Breast Radiotherapy on Acute Toxic Effects of the Skin Among Women With Large Breast Size: A Randomized Clinical Trial. JAMA Oncol. 2022 Jul 1;8(7):994-1000. doi: 10.1001/jamaoncol.2022.1479. PMID 35616948